CLINICAL TRIAL: NCT03638258
Title: A Phase 2b 12-Week Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety, Efficacy and Pharmacokinetics of ARQ-151 Cream 0.3% and ARQ-151 Cream 0.15% Administered Once Daily in Subjects With Chronic Plaque Psoriasis
Brief Title: The Safety, Efficacy and Pharmacokinetics of ARQ-151 Cream in Subjects With Chronic Plaque Psoriasis
Acronym: ARQ-151-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARQ-151-201
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Parallel group, double blind, vehicle-controlled study
Who Masked: Participant, Investigator
Masking Description: Roflumilast drug product will be supplied as a 0.3% and 0.15% cream. The matching vehicle cream will contain only excipients of roflumilast cream.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Roflumilast Cream 0.3% (Experimental): Roflumilast cream 0.3% topically applied QD for 12 weeks.
  Interventions: Drug: Roflumilast Cream 0.3%
- Roflumilast Cream 0.15% (Experimental): Roflumilast cream 0.15% topically applied QD for 12 weeks.
  Interventions: Drug: Roflumilast Cream 0.15%
- Vehicle Cream (Placebo Comparator): Vehicle cream matched to roflumilast cream (containing only excipients of active cream) applied QD for 12 weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.3% — Applied once daily for 12 weeks
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.3%
Drug: Roflumilast Cream 0.15% — Applied once daily for 12 weeks
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.15%
Drug: Vehicle Cream — Applied once daily for 12 weeks
  Arms: Vehicle Cream

SUMMARY:
This is a parallel group, double blind, vehicle-controlled study in which roflumilast (ARQ-151) cream 0.3%, roflumilast cream 0.15%, or vehicle cream is applied once daily (QD) for 84 days to subjects with chronic plaque psoriasis involving between 2 and 20% body surface area.

ELIGIBILITY:
Inclusion Criteria:

* Participants legally competent to sign and give informed consent
* Males and females ages 18 years and older (inclusive)
* Clinical diagnosis of psoriasis vulgaris of at least 6 months duration as determined by the Investigator
* Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at Screening (Visit 1) and Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial.
* In good health as judged by the Investigator, based on medical history, physical examination, serum chemistry labs, hematology values, and urinalysis.
* Subjects are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

* Planned excessive exposure of treated area(s) to either natural or artificial sunlight or tanning bed.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
* Previous treatment with roflumilast cream or its active ingredient
* Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
* Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of study medication.
* Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (30):
- United States (20):
  - Arcutis Clinical Site 35, Beverly Hills, California
  - Arcutis Clinical Site 29, Northridge, California
  - Arcutis Clinical Site 28, San Diego, California
  - Arcutis Clinical Site 27, Santa Monica, California
  - Arcutis Clinical Site 12, Miami, Florida
  - Arcutis Clinical Site 16, Sanford, Florida
  - Arcutis Clinical Site 21, Louisville, Kentucky
  - Arcutis Clinical Site 34, Clinton Township, Michigan
  - Arcutis Clinical Site 33, Detroit, Michigan
  - Arcutis Clinical Site 20, Fridley, Minnesota
  - Arcutis Clinical Site 22, New York, New York
  - Arcutis Clinical Site 14, High Point, North Carolina
  - Arcutis Clinical Site 39, Bexley, Ohio
  - Arcutis Clinical Site 15, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 19, College Station, Texas
  - Arcutis Clinical Site 37, Houston, Texas
  - Arcutis Clinical Site 13, Houston, Texas
  - Arcutis Clinical Site 23, San Antonio, Texas
  - Arcutis Clinical Site 24, Webster, Texas
  - Arcutis Clinical Site 31, Norfolk, Virginia
- Canada (10):
  - Arcutis Clinical Site 18, Surrey, British Columbia
  - Arcutis Clinical Site 11, Surrey, British Columbia
  - Arcutis Clinical Site 38, Winnipeg, Manitoba
  - Arcutis Clinical Site 10, Ajax, Ontario
  - Arcutis Clinical Site 25, London, Ontario
  - Arcutis Clinical Site 26, Markham, Ontario
  - Arcutis Clinical Site 32, Oakville, Ontario
  - Arcutis Clinical Site 17, Peterborough, Ontario
  - Arcutis Clinical Site 30, Waterloo, Ontario
  - Arcutis Clinical Site 36, Windsor, Ontario

REFERENCES:
- [Derived] Stein Gold L, Alonso-Llamazares J, Draelos ZD, Gooderham MJ, Kempers SE, Kircik LH, Lebwohl MG, Papp KA, Pariser DM, Toth DP, Yosipovitch G, Higham RC, Feng A, Berk DR. Effect of Roflumilast Cream (ARQ-151) on Itch and Itch-Related Sleep Loss in Adults with Chronic Plaque Psoriasis: Patient-Reported Itch Outcomes of a Phase 2b Trial. Am J Clin Dermatol. 2023 Mar;24(2):305-313. doi: 10.1007/s40257-022-00739-3. Epub 2022 Nov 12. PMID 36370336
- [Derived] Lebwohl MG, Papp KA, Stein Gold L, Gooderham MJ, Kircik LH, Draelos ZD, Kempers SE, Zirwas M, Smith K, Osborne DW, Trotman ML, Navale L, Merritt C, Berk DR, Welgus H; ARQ-151 201 Study Investigators. Trial of Roflumilast Cream for Chronic Plaque Psoriasis. N Engl J Med. 2020 Jul 16;383(3):229-239. doi: 10.1056/NEJMoa2000073. PMID 32668113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (≥18 years of age) male or female participants with chronic plaque psoriasis were recruited at 30 study sites in the US and Canada.
Groups:
- Rolumilast Cream 0.3%: Roflumilast (ARQ-151) cream 0.3% was topically applied once daily (QD) for 12 weeks.
- Roflumilast Cream 0.15%: Roflumilast (ARQ-151) cream 0.15% was topically applied QD for 12 weeks.
- Vehicle Cream: Vehicle cream matched to roflumilast cream (containing only excipients of active cream) was applied topically QD for 12 weeks.
Period: Overall Study
Arm/Group | Rolumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Started | 109 | 113 | 109
Completed | 102 | 104 | 86
Not Completed | 7 | 9 | 23
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 4 | 5
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5 | 12
Not completed — Lack of Efficacy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Roflumilast Cream 0.3%: Roflumilast cream 0.3% was topically applied QD for 12 weeks.
- Roflumilast Cream 0.15%: Roflumilast cream 0.15% was topically applied QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total
Number analyzed (Participants) | 109 | 113 | 109 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.11) | 54.4 (14.20) | 55.5 (13.49) | 53.9 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 42 | 146
  Male | 56 | 62 | 67 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 26 | 25 | 76
  Not Hispanic or Latino | 84 | 87 | 84 | 255
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 8 | 7 | 5 | 20
  Native Hawaiian or Other Pacific Islander | 12 | 10 | 7 | 29
  Black or African American | 0 | 0 | 0 | 0
  White | 82 | 95 | 92 | 269
  More than one race | 7 | 1 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Whole Body Investigator Global Assessment (IGA) Score [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
  Participants
    0 - Clear | 0 | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0 | 0
    2 - Mild | 17 | 18 | 11 | 46
    3 - Moderate | 84 | 83 | 89 | 256
    4 - Severe | 8 | 12 | 9 | 29
Intertriginous Area Investigator Global Assessment (I-IGA) Score [Count of Participants; unit: Participants] — The I-IGA is 5-point scale assessing the severity of plaque psoriasis in the intertriginous area, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity. Population: All randomized participants with intertriginous area involvement are included.
  Participants
    1 - Almost Clear: number analyzed (Participants) | 16 | 18 | 17 | 51
    1 - Almost Clear | 1 | 2 | 0 | 3
    2 - Mild: number analyzed (Participants) | 16 | 18 | 17 | 51
    2 - Mild | 6 | 12 | 7 | 25
    3 - Moderate: number analyzed (Participants) | 16 | 18 | 17 | 51
    3 - Moderate | 8 | 3 | 8 | 19
    4 - Severe: number analyzed (Participants) | 16 | 18 | 17 | 51
    4 - Severe | 1 | 1 | 2 | 4
Itch-Related Sleep Loss Score [Mean (Standard Deviation); unit: score on a scale] — The Itch-Related Sleep Loss NRS is a single item scale scored from 0 ("no itch-related sleep loss") to 10 ("itch-related sleep loss as bad as it could be") assessing the severity of itch-related sleep loss in the past 24 hours. Higher scores indicate greater symptom severity.
  score on a scale | 2.9 (3.24) | 3.0 (3.19) | 3.4 (3.18) | 3.1 (3.20)
Percentage of Body Surface Area (BSA) Affected [Mean (Standard Deviation); unit: percentage of body surface area] | 6.33 (4.005) | 6.44 (3.915) | 6.43 (3.597) | 6.40 (3.833)
Modified Psoriasis Area Severity Index (mPASI) Score [Mean (Standard Deviation); unit: score on a scale] — The mPASI combines assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity. The body is divided into four sections (head (h) (10% of a person's skin); arms (a) (20%); trunk (t) (30%); legs (l) (40%)). Each of these areas is scored alone, and then the four scores are combined into the final mPASI. For each section, the percent of area (A) of skin involved is estimated and then transformed into a grade from 0 ("0% of area involved") to 6 ("90 to 100% of involved area").
  score on a scale | 5.94 (3.959) | 6.33 (4.363) | 5.77 (3.498) | 6.02 (3.956)
Worst Itch - Numerical Rating Scale (WI-NRS) Score [Mean (Standard Deviation); unit: score on a scale] | 6.1 (2.67) | 5.6 (3.05) | 5.9 (2.87) | 5.9 (2.87)
Total Psoriasis Symptom Diary (PSD) Score [Mean (Standard Deviation); unit: score on a scale] | 68.9 (41.18) | 69.6 (46.20) | 75.1 (42.55) | 71.2 (43.35)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: score on a scale] | 6.7 (5.50) | 8.8 (7.15) | 8.5 (5.62) | 8.0 (6.17)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' at Week 6
Description: The percentage of participants with an IGA score of 0 ('clear') or 1 ('almost clear') at Week 6 is reported. The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
Time Frame: Week 6
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Groups:
- Vehicle Cream: Vehicle cream matched to roflumilast cream (containing only excipients of ARQ-151 cream) was applied topically QD for 12 weeks.
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants | 28.0 | 22.8 | 8.3
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Test type: Superiority — Missing data imputed using linear interpolation and last observation carried forward (LOCF) where linear interpolation was not computationally possible; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpolation was not computationally possible; p = 0.004, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score

2. Secondary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear'
Description: The percentage of participants with an IGA score of 0 ('clear') or 1 ('almost clear') is reported. The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
Time Frame: Weeks 4, 8, and 12
Population: All randomized participants are included. Missing data from subjects was handled with linear interpolation (subjects with assessments before and after the missing assessment) or last observation carried forward (LOCF) [subjects with assessments only before the missing assessment].
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | 14.5 | 9.0 | 4.4
  Week 8 | 37.9 | 30.6 | 11.9
  Week 12 | 37.5 | 32.1 | 16.3
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and last observation carried forward where linear interpolation was not computationally possible; p = 0.015, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from placebo at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.174, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.008, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score

3. Secondary Outcome: Change From Baseline in Modified Psoriasis Area Severity Index (mPASI) Score
Description: The percent change from baseline in mPASI score is presented. The mPASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity. For scoring, the body is divided into four sections (head [h]: 10% of a person's skin; arms [a] 20%; trunk [t] 30%; legs (l] 40%); for each section, the percent of area involved is estimated from 0 (0% involved) to 6 (90 to 100% involved). Then, within each area, the severity is estimated by three clinical signs: erythema ('E'; redness), induration ('T'; thickness), and desquamation ('S'; scaling). Severity parameters are measured on a scale of 0 to 4, from none to maximum severity possible. Each of these areas is scored by itself, and then the four scores are combined into the final mPASI, using the formula mPASI = 0.1 (Eh + Th + Sh) Ah + 0.2 (Ea + Ta + Sa) Aa + 0.3 (Et + Tt + St) At + 0.4 (El + Tl + Sl) Al.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: All randomized participants are included. Missing data from subjects was handled with linear interpolation (subjects with assessments before and after the missing assessment) or LOCF (subjects with assessments only before the missing assessment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
score on a scale
  Week 4 | -40.08 (46.811) | -47.32 (29.717) | -18.01 (46.622)
  Week 6 | -53.15 (46.470) | -59.73 (32.409) | -16.42 (58.385)
  Week 8 | -59.09 (49.290) | -65.12 (31.97) | -18.47 (63.777)
  Week 12 | -59.48 (54.881) | -68.03 (33.021) | -13.65 (70.731)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15%; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible.x; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline mPASI score

4. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) Affected
Description: The BSA affected by psoriasis was determined by the subject's hand method, where the subject's hand (including fingers) surface area was assumed to equal 1% of BSA. The mean percent change from baseline in BSA is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of change
  Week 4 | -21.74 (34.381) | -23.25 (27.084) | -5.33 (31.834)
  Week 6 | -34.88 (39.530) | -33.41 (32.136) | -8.19 (40.989)
  Week 8 | -41.58 (42.816) | -40.49 (34.379) | -7.40 (52.859)
  Week 12 | -48.56 (46.077) | -47.50 (36.304) | -6.74 (51.469)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream on Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline BSA score

5. Secondary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear' Plus a 2-Grade Improvement From Baseline
Description: The percentage of participants with an IGA score of 0 ('clear') or 1 ('almost clear') plus a 2-grade improvement from baseline is reported. The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | 10.0 | 6.9 | 4.4
  Week 6 | 23.9 | 17.4 | 8.0
  Week 8 | 32.2 | 24.5 | 9.8
  Week 12 | 31.3 | 27.4 | 13.6
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.116, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.423, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.002, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.038, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.005, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.002, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.013, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline IGA score

6. Secondary Outcome: Percentage of Participants With an Intertriginous Area Investigator Global Assessment (I-IGA) Score of 'Clear' or 'Almost Clear' Who Had at Least Mild Lesions at Baseline
Description: The percentage of participants (who had intertriginous area involvement with an I-IGA score of at least mild at baseline) with at least a 2-grade improvement in I-IGA score at Weeks 4, 6, 8, and 12 is presented.
Time Frame: Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | 46.6 | 43.8 | 17.6
  Week 6 | 73.4 | 43.7 | 29.4
  Week 8 | 87.1 | 60.9 | 36.1
  Week 12 | 94.3 | 32.4 | 24.3
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference form vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.086, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.123, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.017, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.415, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.007, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.175, Regression, Linear; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.619, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline I-IGA score

7. Secondary Outcome: Change From Baseline in Worst Itch-Numeric Rating Scale (WI-NRS) Pruritus Score
Description: The WI-NRS is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. The mean (SD) change in WI-NRS score from baseline is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
score on a scale
  Week 4 | -2.8 (2.53) | -1.9 (2.45) | -1.1 (2.20)
  Week 6 | -3.3 (2.56) | -2.6 (2.73) | -1.3 (2.67)
  Week 8 | -3.5 (2.59) | -2.9 (2.73) | -1.5 (3.00)
  Week 12 | -3.4 (2.76) | -3.2 (2.84) | -1.3 (2.76)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.002, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score

8. Secondary Outcome: Percentage of Participants With Baseline Worst Itch-Numeric Rating Scale (WI-NRS) Pruritus Score ≥6 Who Experienced a 4-point Reduction
Description: The percentage of participants who had baseline WI-NRS scores ≥6 who achieved a 4-point reduction in WI-NRS score at Weeks 4, 6, 8, and 12 is reported. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: All randomized participants with a WI-NRS score ≥6 at baseline are included. All randomized participants are included. Missing data from subjects was handled with linear interpolation (subjects with assessments before and after the missing assessment) or LOCF (subjects with assessments only before the missing assessment).
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 71 | 62 | 64
percentage of participants
  Week 4 | 50.9 | 35.4 | 24.9
  Week 6 | 52.8 | 57.0 | 34.5
  Week 8 | 64.6 | 58.2 | 42.3
  Week 12 | 62.8 | 70.1 | 32.9
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.002, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.203, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.034, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.012, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.010, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.075, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, Regression, Logistic; Logistic regression with a factor of treatment group and a covariate of baseline WI-NRS score

9. Secondary Outcome: Percentage of Participants Achieving a Modified Psoriasis Area Severity Index-75 (mPASI-75) Compared to Baseline
Description: The percentage of subjects achieving a 75% reduction in mPASI (eg, mPASI-75) score relative to baseline is presented. The mPASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | 13.3 | 7.6 | 10.5
  Week 6 | 24.1 | 22.2 | 9.6
  Week 8 | 31.3 | 23.0 | 13.2
  Week 12 | 34.1 | 31.1 | 16.0
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.527, Regression, Logistic; Logistic regression (Firth's penalized likelihood) with a factor of treatment group and a covariate of baseline PASI score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.444, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.006, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.013, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.002, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.064, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.002, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.009, Regression, Logistic; [statistical method as in outcome 9, analysis 1]

10. Secondary Outcome: Percentage of Participants Achieving a Modified Psoriasis Area Severity Index-90 (mPASI-90) Compared to Baseline
Description: The mPASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity. The percentage of subjects achieving a 90% reduction in mPASI (eg, mPASI-90) score relative to baseline is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | 6.0 | 1.3 | 2.3
  Week 6 | 14.3 | 2.3 | 3.2
  Week 8 | 16.9 | 7.4 | 6.0
  Week 12 | 20.6 | 13.7 | 7.8
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.188, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.577, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.008, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.664, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.015, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.666, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.009, Regression, Logistic; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.163, Regression, Logistic; [statistical method as in outcome 9, analysis 1]

11. Secondary Outcome: Change From Baseline in Psoriasis Symptom Diary (PSD) Total Score
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 11 ("worst imaginable symptoms"). Scores range from 0 to 176, with higher scores indicating greater symptom severity. The mean (SD) change in PSD total score relative to baseline is presented for each treatment arm.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
percentage of participants
  Week 4 | -32.7 (34.61) | -32.7 (35.08) | -22.9 (31.85)
  Week 6 | -37.8 (35.71) | -38.0 (37.88) | -24.6 (38.15)
  Week 8 | -40.5 (36.62) | -40.1 (39.04) | -26.9 (41.78)
  Week 12 | -40.8 (41.12) | -43.4 (40.44) | -23.0 (41.38)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream on Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible. ANCOVA with a factor of treatment group and a covariate of baseline PSD score; p = 0.002, ANOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.002, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from placebo at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from placebo at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline PSD score

12. Secondary Outcome: Change From Baseline in Itch-Related Sleep Loss Numeric Rating Scale (NRS) Score
Description: The Itch-Related Sleep Loss NRS is a single item scale scored from 0 ("no itch-related sleep loss") to 10 ("itch-related sleep loss as bad as it could be") assessing the severity of itch-related sleep loss in the past 24 hours. The mean (SD) change from the baseline NRS score is presented for each treatment arm.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
score on a scale
  Week 4 | -1.1 (2.95) | -1.2 (2.54) | -1.0 (2.74)
  Week 6 | -1.5 (2.94) | -1.3 (2.65) | -0.9 (2.96)
  Week 8 | -1.6 (2.96) | -1.7 (2.75) | -0.9 (3.08)
  Week 12 | -1.8 (3.01) | -1.7 (2.66) | -1.1 (3.33)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.184, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from placebo at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.207, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.004, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.022, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.003, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p < 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible. ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score; p = 0.003, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.01, ANCOVA — ANCOVA with a factor of treatment group and a covariate of baseline Itch-Related Sleep Loss NRS score

13. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a 10-item scale asking subject to rate the severity of symptoms during the past week. Each item is scored from 0 ("not at all" or "not relevant") to 3 or 4 ("very much") [2 questions are scored 0 to 3 and 8 questions are scored 0 to 4]. The total DLQI score ranges from 0 to 48, with higher scores indicating greater symptom severity. The mean (SD) change from baseline DLQI score is presented.
Time Frame: Baseline (Day 1) and Weeks 4, 6, 8, and 12
Population: This endpoint was added in protocol amendment 1. All participants randomized after implementing amendment 1 are included. All randomized participants are included. Missing data from subjects was handled with linear interpolation (subjects with assessments before and after the missing assessment) or LOCF (subjects with assessments only before the missing assessment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 58 | 60 | 62
score on a scale
  Week 4 | -2.2 (3.46) | -2.3 (4.01) | -1.9 (4.29)
  Week 6 | -2.6 (3.64) | -3.1 (4.23) | -1.8 (4.23)
  Week 8 | -2.6 (3.68) | -3.5 (4.57) | -1.6 (4.77)
  Week 12 | -2.6 (4.48) | -4.2 (4.92) | -1.4 (5.28)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.255, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream on Week 4; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.687, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.045, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 6; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.059, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 5: Comparison: Roflumilast Cream 0.3%; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.051, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 8; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.013, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 7: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.036, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score
Statistical Analysis 8: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Difference from vehicle cream at Week 12; Test type: Superiority — Missing data imputed using linear interpolation and LOCF where linear interpretation was not computationally possible; p = 0.001, ANCOVA; ANCOVA with a factor of treatment group and a covariate of baseline DLQI score

14. Secondary Outcome: Responses to Individual Questions of the Psoriasis Symptom Diary (PSD)
Description: Two items from the PSD asking participants to rate the overall severity of psoriasis-related itching and pain during the past 24 hours are presented. Each item is scored on an 11-point scale ranging from 0 ("no symptom") to 10 ("worst imaginable symptom"), with lower scores indicating lower symptoms severity. The mean (SD) score is presented for each treatment arm.
Time Frame: Weeks 4, 6, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 109 | 113 | 109
score on a scale
  Week 4: Itching | 3.0 (2.87) | 3.3 (2.88) | 4.2 (3.02)
  Week 4: Pain | 1.8 (2.67) | 1.6 (2.46) | 2.6 (2.89)
  Week 6: Itching | 2.7 (2.70) | 2.8 (2.80) | 4.2 (2.96)
  Week 6: Pain | 1.5 (2.39) | 1.5 (2.52) | 2.3 (2.70)
  Week 8: Itching | 2.4 (2.70) | 2.4 (2.69) | 4.0 (2.92)
  Week 8: Pain | 1.3 (2.48) | 1.3 (2.36) | 2.4 (2.76)
  Week 12: Itching | 2.3 (2.78) | 2.2 (2.65) | 4.3 (3.14)
  Week 12: Pain | 1.2 (2.37) | 1.2 (2.35) | 2.5 (2.94)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: All enrolled participants are included in analysis of all-cause mortality. All participants who received ≥1 dose of study therapy are included in analysis of serious adverse events (SAEs) and nonserious adverse events (AEs).
Arm/Group | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/113 | 0/109
Serious Adverse Events (participants affected / at risk) | 1/109 | 1/110 | 2/107
Other Adverse Events (participants affected / at risk) | 8/109 | 7/110 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.3% (N=109) | Roflumilast Cream 0.15% (N=110) | Vehicle Cream (N=107)
Chest pain (Cardiac disorders) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal ganglia infarct (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.3% (N=109) | Roflumilast Cream 0.15% (N=110) | Vehicle Cream (N=107)
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT03638258/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03638258/SAP_002.pdf